CLINICAL TRIAL: NCT07382609
Title: The Effect of Creating a Birth Story in the Labor Room on Fear of Childbirth and Birth Comfort in Primiparous Pregnant Women
Brief Title: The Effect of Creating a Birth Story in the Labor Room on Fear of Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra Tan, Master's Degree Student in Midwifery, Clinical Midwife, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5499
Record Dates: First submitted 2024-12-09; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Birth
Keywords: comfort; fear of birth; pregnant

STUDY DESIGN:
Intervention Model Description: Crossover Assignment randomized controlled trial conducted with experimental and control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: (No Intervention): GROUP WITHOUT BIRTH STORY
- Experimental (Experimental): Birth story creating group
  Interventions: Behavioral: BIRTH STORY EXPERIMENTAL GROUP

INTERVENTIONS:
Behavioral: BIRTH STORY EXPERIMENTAL GROUP — The birth story is created by the pregnant women in the labor room writing their feelings on a transparent wallpaper attached to the wall. The pregnant woman, the midwife, the father and the doctor can also write their feelings and thoughts on this wallpaper. In this way, the pregnant woman looks at the wall on which positive thoughts are written throughout the labor and thus the fear of birth is reduced.
  Arms: Experimental

SUMMARY:
The aim of this study is to reduce the fears of women who will give birth and increase their comfort. In the literature review conducted for this purpose, no study has yet been found that examines the effect of creating a birth story in the labor room on the fear of birth and birth comfort in primiparous pregnant women. In order to fill this gap in the literature, pregnant women in the labor room will be asked to create their birth stories and the effect of this on fear of birth and birth comfort will be examined.

The hypotheses of the study are as follows:

H1a: Creating a birth story in the labor room affects fear of birth H1b: Creating a birth story in the labor room affects birth comfort.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of creating a birth story in the labor room on the fear of childbirth and the comfort of pregnant women. Data will be collected from primiparous pregnant women who are admitted to the labor room in the maternity ward of Gölbaşı State Hospital and are in the latent phase. Women will be informed about the study and will be asked whether they will participate in the study. Informed consent forms will be distributed to women who agree to participate in the study. Data collection tools will be applied to women who agree to participate in the study by the researcher through face-to-face interviews. Data collection will be completed with the end of the latent phase (≥ 4-6 cm). No intervention will be applied to women in the control group, however, the Personal Information Form, Prenatal Self-Assessment Scale-Fear of Childbirth Subscale and Childbirth Comfort Scale will be applied simultaneously with the experimental group. Pre-test data collection questionnaires will be applied to pregnant women in the experimental group at the beginning of the latent phase and pregnant women will be asked to create their own birth stories. A transparent wall board will be attached to the wall of the labor room and pregnant women will be given appropriate pens and asked to write their feelings and thoughts on this board and in this way, birth stories will be created. If pregnant women wish, their photographs will be taken and attached to this board. After the birth story is created, the post-test data collection tools will be applied to the pregnant woman again and the data collection process will be completed.

ELIGIBILITY:
Inclusion Criteria:- All primiparous pregnant women who are literate,

* Over the age of 18,
* Not experiencing a risky pregnancy,
* Not becoming pregnant with assisted reproductive techniques,
* Planned to have a vaginal birth,
* In the latent phase of labor,
* Do not have any psychiatric disorders,
* Do not have any health problems in themselves or their babies,
* Do not have a history of ex fetus will be included in the study.

Exclusion Criteria:

* Pregnant women with an indication for caesarean section during the latent phase of labour will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 58 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Prenatal Self Evaluation Questionnaire score | Baseline (latent phase of labor) and prior to active labor (at 4 cm cervical dilatation)]
  The scale developed by Lederman determines women's adaptation to pregnancy and motherhood. This scale is a 4-point Likert-type scale with 7 sub-dimensions and 79 items. The scores that can be obtained from the scale are between 10 and 40.

SECONDARY OUTCOMES:
Childbirth Comfort Questionnaire- CCQ score | Immediately prior to active labor (at 4 cm cervical dilatation)
  The scale consists of 9 questions and is a 5-point Likert type (1=Strongly disagree, 2=Mostly disagree, 3=Partially agree, 4=Mostly agree, 5=Totally agree). The items are expected to be answered considering the comfort of the delivery room. Each statement reports a certain sense of comfort (relaxation, relief or superiority) and dimensions (physical, environmental, psychospiritual or social). A minimum of 9 and a maximum of 45 points can be obtained from the scale. It can be thought that as the score value of the scale increases, comfort increases, and as the score value decreases, comfort decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Esra GÜNEY, PhD, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Battalgazi̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research results will be shared.

REFERENCES:
- See also: Description Reference link — https://pubmed.ncbi.nlm.nih.gov/39568156/